CLINICAL TRIAL: NCT06941064
Title: Relating Anthropometric Profile and Countermovement Jump Performance to In-Match GPS-Derived External Load Metrics in Mexican National Team Soccer Players
Brief Title: Relationship of Anthropometric Profile and Fitness Indicators With Sports Performance of Elite Mexican National Team Soccer Players
Acronym: ANTHROPERFORMX
Status: Enrolling by invitation | Type: Observational
Sponsor: Iberoamerican Institute of Sports Science and Human Movement (Other)
Collaborators: Metropolitan Autonomous University (Other)
Responsible Party: Principal Investigator, Cesar Octavio Ramos Garcia, PhD, Pricnipal investigator, Iberoamerican Institute of Sports Science and Human Movement
Other Study IDs: FMF-IICDEM-ID-001-2025
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Athletes; Soccer
Keywords: Kinanthropometry; Body Composition; Sports Performance; Somatotype
MeSH Terms: interventions — Body Composition; Anthropometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elite Mexican soccer players: Mexican National Team soccer players gathered at the Mexican Football Federation facilities before official international matches will be considered to participate in the study.
  Interventions: Diagnostic Test: Anthropometric and sports performance assessment

INTERVENTIONS:
Diagnostic Test: Anthropometric and sports performance assessment — According to the International Society for the Advancement of Kinanthropometry (ISAK) standards, sixteen anthropometric variables have been assessed to characterize the athlete's anthropometric profile. The counter-movement jump assessments were conducted using a ForceDecks Max platform. During matches, the players' GPS-derived external Load Metrics were monitored using 18 Hz WIMU Pro GPS units. Normality tests of all variables will be performed.
  Certificated anthropometrists performed the anthropometric assessment twice. A third measurement will be performed if the difference between these measures exceeds 5% for skinfolds and 1% for all other variables. Countermovement jump tests were conducted in duplicate, and the higher measurements were recorded. In-match GPS-derived external load metrics of different matches will be downloaded and analyzed.
  Other Names: Body composition; Anthropometry; Fitness; Sports Performance

SUMMARY:
Relating Anthropometric Profile to Fitness and Sports Performance in Mexican National Team Soccer Players

DETAILED DESCRIPTION:
Previous studies have reported differences in the body composition of Latin American or European youth to elite soccer players based on playing position or age. Furthermore, in youth or sub-elite samples, body composition has been linked to in-match speed, distance, or acceleration. Few studies have been developed with elite samples of soccer players. Elite soccer performance depends on the complex interaction of physical, physiological, tactical, and contextual variables. Therefore, a comprehensive analysis of anthropometric, countermovement jump and in-match performance variables can provide deeper insight into soccer success. Accordingly, this study addresses this knowledge gap by characterizing and analyzing the multidimensional relationships between these variables in elite Mexican soccer players. A descriptive, cross-sectional study will be conducted. According to the International Society for the Advancement of Kinanthropometry (ISAK) standards, sixteen anthropometric variables have been assessed to characterize the athlete's anthropometric profile. The counter-movement jump assessments were conducted using a ForceDecks Max platform. During matches, the players' displacement was monitored using 18 Hz WIMU Pro GPS units. Normality tests of all variables will be performed. A descriptive analysis of anthropometric and body composition characteristics of overall and among playing positions will be performed. The relationship between body composition and anthropometric profile with counter-movement jump and in-match GPS-Derived External Load Metrics will be computed. Multivariate models will be explored to analyze multidimensional relationships between these variables.

ELIGIBILITY:
Inclusion Criteria:

* Athletes who attended the evaluation laboratories.
* Athletes who gave their assent to carry out the evaluations.
* Female or male soccer players.
* Actively competing in national and/or international tournaments.

Exclusion Criteria:

* Not having been called to integrate the Mexican national soccer team during the evaluation dates.
* Injured or ill athletes during the assessments.
* Athletes who do not give their assent to carry out the evaluations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mexican National Team soccer players gathered at the Mexican Football Federation facilities before official international matches.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-07-11 (Estimated); Study Completion 2025-12-11 (Estimated)

PRIMARY OUTCOMES:
Anthropometric profile | One day
  Anthropometric assessment through the International Society for the Advancement in Kinanthropometry standards

SECONDARY OUTCOMES:
Countermovement jump performance | One day
  An assessment of lower-limb strength and power using ForceDecks Max platform (VALD Performance, Australia).
GPS-derived external load metrics | One day
  In-match players' sports performance will be monitored during matches using 18 Hz WIMU Pro GPS units (RealTrack Systems, Almería, Spain).

CONTACTS AND LOCATIONS:
Overall Officials: William Carvajal Veitía, Principal Investigator — Institute of Sports Medicine, Cuba; Rodrigo Yáñez Sepúlveda, Principal Investigator — Andres Bello University (UNAB), Chile; Luis Ortíz Hernández, Principal Investigator — Metropolitan Autonomous University campus Xochimilco; Israel Rios Limas, Principal Investigator — Mexican Football Federation; Andrés López Sagarra, Principal Investigator — Mexican Football Federation; José F López Gil, Principal Investigator — Universidad de las Américas (UDLA), Ecuador
Locations (1):
- Mexican Football Federation, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
Because the participants were informed that data management would be protected only by the principal investigators.

REFERENCES:
- [Background] Ju W, Cost R, Oliva-Lozano JM. Analysis of match performance of elite soccer players across confederations during the Men's and Women's World Cup. Sci Med Footb. 2025 Nov;9(4):369-381. doi: 10.1080/24733938.2024.2409679. Epub 2024 Sep 30. PMID 39347689
- [Background] Carlos-Vivas J, Franco-Garcia JM, Mendoza-Munoz DM, Gomez-Pomares S, Perez-Gomez J. High-Intensity GPS-Derived Parameters in Semi-Professional Soccer: Home vs. Away Roles of the Team and Their Relationship with the Match's Final Score. Sensors (Basel). 2024 Jul 27;24(15):4891. doi: 10.3390/s24154891. PMID 39123938
- [Background] Ramirez-Munera M, Arcusa R, Lopez-Roman FJ, Avila-Gandia V, Perez-Pinero S, Munoz-Carrillo JC, Luque-Rubia AJ, Marhuenda J. Relationship Between Anthropometric Profile, Body Composition, and Physical Performance in Spanish Professional Female Soccer Players at Pre-Season Onset: A Cross-Sectional Study. J Funct Morphol Kinesiol. 2025 Feb 27;10(1):79. doi: 10.3390/jfmk10010079. PMID 40137331
- [Background] Ishida A, Travis SK, Stone MH. Associations of Body Composition, Maximum Strength, Power Characteristics with Sprinting, Jumping, and Intermittent Endurance Performance in Male Intercollegiate Soccer Players. J Funct Morphol Kinesiol. 2021 Jan 7;6(1):7. doi: 10.3390/jfmk6010007. PMID 33462168
- [Background] Petri C, Campa F, Holway F, Pengue L, Arrones LS. ISAK-Based Anthropometric Standards for Elite Male and Female Soccer Players. Sports (Basel). 2024 Feb 23;12(3):69. doi: 10.3390/sports12030069. PMID 38535732
- [Background] Radziminski L, Szwarc A, Padron-Cabo A, Jastrzebski Z. Correlations between body composition, aerobic capacity, speed and distance covered among professional soccer players during official matches. J Sports Med Phys Fitness. 2020 Feb;60(2):257-262. doi: 10.23736/S0022-4707.19.09979-1. Epub 2019 Oct 24. PMID 31663315